CLINICAL TRIAL: NCT04584294
Title: MyPath: A Patient-Centered Web-Based Intervention to Improve Reproductive Planning for Women Veterans
Brief Title: Patient-Centered Reproductive Decision Support Tool for Women Veterans
Acronym: MyPath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Kaiser Permanente (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 19-387
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Contraception; Contraception Behavior; Prepregnancy Health; Reproductive Health
Keywords: Shared decision making; Primary care; Patient decision support; Patient-centered outcomes research; Reproductive autonomy; Patient-Centered Care; Provider-Patient Communication
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: Provider participants are randomized to one of two groups - usual care or intervention group - at the start of the study, prior to any Veteran enrollment. Subsequently, Veterans scheduled to see these providers will be enrolled as patient participants and automatically allocated to the study group of their scheduled provider.
Who Masked: Outcomes Assessor
Masking Description: Research assistants (RAs) who assess outcomes will remain blinded to provider study arm assignment throughout the trial. RAs will be blinded to patient study arm assignment during patient enrollment and baseline surveys but will become unblinded to individual patient study arm assignment during the course of outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (MyPath) (Experimental): Patients scheduled to see providers randomized to this arm will receive a weblink to the decision tool via text message after study enrollment and prior to their scheduled visit.
  Interventions: Behavioral: MyPath Web-Based Informational and Decision Support Tool
- Usual Care (No Intervention): Patients scheduled to see providers randomized to the usual care arm will receive no intervention and will receive usual primary care.

INTERVENTIONS:
Behavioral: MyPath Web-Based Informational and Decision Support Tool — The MyPath Decision Support Tool includes the following sections and features:
  * Questions to capture reproductive goals and orientations towards a potential pregnancy
  * Education modules about the menstrual cycle, fertility, and prepregnancy health with the opportunity to flag topics that are relevant and of interest to the patient
  * A contraceptive decision module that provides education, elicits patient preferences about different aspects of contraception, and suggests methods most appropriate based on the patient's preferences
  * A feature for adding free-text questions that patients may have for their provider
  * An email with a summary page that the patient can bring to a visit to guide discussions with primary care providers about reproductive needs
  Arms: Intervention (MyPath)

SUMMARY:
The investigators have developed a web-based decision support tool to help women Veterans get the information and care they need to achieve their reproductive goals, whether that includes optimizing their health before desired pregnancies or birth control to avoid unwanted pregnancies. The study will test the effect of sending a weblink to the decision tool to women Veterans prior to primary care visits at the VA. Half of participants will be sent a weblink before their appointment, and half will not be sent the link. The investigators hypothesize that participants who are sent the link will be more likely to report patient-centered discussions of their reproductive needs at visits, feel confident in communicating with their health care providers, have accurate knowledge about reproductive health, and choose birth control methods that best fit their preferences and needs.

DETAILED DESCRIPTION:
Counseling and care that supports individuals' ability to achieve their reproductive goals is an essential component of primary care. National organizations, including the Centers for Disease Control and Prevention (CDC), recommend that clinicians routinely engage in patient-centered conversations about reproductive goals and offer care to help optimize health and well-being prior to desired pregnancies and to prevent unwanted pregnancy and births. This counseling is particularly critical for women Veterans, who face elevated risks of adverse pregnancy and birth outcomes due to a high prevalence of chronic medical and mental health conditions as well as psychosocial stressors including sexual trauma histories, intimate partner violence, and homelessness. Moreover, stark racial/ethnic disparities in pregnancy outcomes are well-documented, and nearly half of reproductive-aged women Veterans are minority race/ethnicity. Despite these national recommendations, however, conversations about reproductive needs are often absent in primary care both outside and within the VA, and the conversations that do happen frequently fail to incorporate women's values and preferences. Interventions are needed to improve both the frequency and quality of counseling about reproductive needs in primary care settings.

This study will investigate the effect of a novel, web-based, patient-facing decision support tool designed to be used prior to VA primary care visits to help women Veterans with reproductive capacity consider their reproductive goals; improve their knowledge about fertility, contraception, and prepregnancy health risks; align contraceptive decisions with their preferences and goals; and engage in shared decision making (SDM) with providers.

The investigators will conduct a multi-site randomized controlled trial (RCT) clustered at the provider level among VA primary care providers and their reproductive-aged women Veteran patients. Study outcomes will be assessed among participants shortly after their scheduled appointment and at 3- and 6-months follow up. The study will test the primary hypothesis that participants who receive the tool weblink prior to visits will be more likely to report patient-centered conversations about their reproductive needs at their visit. The investigators also hypothesize that intervention participants will report higher perceived self-efficacy in communicating with providers, reproductive health knowledge, contraception decision quality, and contraception utilization. Exploratory outcomes include behaviors to modify preconception health risks among participants considering pregnancy in the future and intervention effects by race/ethnicity. The study will also collect quantitative and qualitative data to assess the feasibility of implementing the tool more widely in VA primary care settings.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Female sex identified in medical record
* 18 - 44 years old
* Has a scheduled VA medical appointment with an enrolled study provider
* Has at least one valid telephone number available in medical record
* Interested in receiving information or talking with their provider about pregnancy and/or birth control

Providers:

* Primary Care Provider (MD, Nurse Practitioner, Physician Assistant) at a study site
* Designated as a Women's Health Provider [defined in VA directive 1330.01 as primary care providers who have demonstrated proficiency (e.g. pelvic exams and pap smears) in women's health and who have at least 10% of their panel comprised of women]
* Completed appointments with at least 30 unique female patients ages 18-44 in the past year at a study site

Exclusion Criteria:

Patients:

* Currently pregnant
* Medical record or self-reported history of hysterectomy, bilateral oophorectomy; or self-report of not having a uterus
* Unable to communicate in English
* Impaired decision-making
* Used the decision tool prior to study enrollment (e.g. during pilot testing of the tool)

Providers:

* Previous involvement as a provider in MyPath pilot work (identified by the PI)
* Medical trainee
* Self-report that they have plans to leave VA, go on extended leave, retire, stop primary care practice, or change VA site in the 18 months following their enrollment

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 465 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S Callegari, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (12):
- United States (12):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Orlando VA Medical Center, Orlando, FL, Orlando, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - El Paso VA Health Care System, El Paso, TX, El Paso, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - Central Texas Veterans Health Care System, Temple, TX, Temple, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Veteran participant data will be deposited into the "Reproductive, Sexual, and Socio-Behavioral Health Data Repository and Registry" VA data repository and registry housed and managed at the VA Puget Sound Health Care System. The data will be stored indefinitely in accordance with VHA regulations under VA IRB and R&D Committee oversight. Procedures are as follows.
Time Frame: Data will be deposited into the data repository and registry described above at study closure. It is the intention of the repository team to store the data in the repository indefinitely.
  In accordance with VHA regulations, the repository will be terminated only under the direction of the VA IRB or R&D Committee responsible for the oversight of the repository. If the repository is terminated, the data will only be re-used or transferred to another data repository if the IRB and/or R&D approves of the transfer. The repository data may need to be destroyed if appropriate control of the data and compliance with VA and VHA requirements cannot be maintained.
  If the repository is terminated, the data will be destroyed in accordance with all VA and VHA records disposition requirements. We will retain these data for the minimum period required for records retention in accordance with the National Archives and Records Administration (NARA) VHA Record Control Schedule (RCS).
Access Criteria: Study data may be requested by VA investigators (all investigators must receive regulatory approval and sign a Data Use Agreement before gaining access to the data). The data repository will only be used to answer questions for approved studies and/or for activities preparatory to research. For activities preparatory to research, staff may only use aggregate data, and only for background information, to justify the research, or to verify proposed sample size requirements.
  Data from this study will be made available outside VA in response to a properly prepared Freedom of Information Act request submitted to the VA Puget Sound FOIA Officer, or submitted and passed down to the facility FOIA Officer from higher VA authority (e.g. VISN 20 or Central Office). Research publications will be made available to the public via the National Library of Medicine PubMed Central website within one year after publication date(s).

REFERENCES:
- [Result] Callegari LS, Benson SK, Mahorter SS, Nelson KM, Arterburn DE, Hamilton AB, Taylor L, Hunter-Merrill R, Gawron LM, Dehlendorf C, Borrero S. Evaluating the MyPath web-based reproductive decision support tool in VA primary care: Protocol for a pragmatic cluster randomized trial. Contemp Clin Trials. 2022 Nov;122:106940. doi: 10.1016/j.cct.2022.106940. Epub 2022 Sep 28. PMID 36179982

RESULTS

PARTICIPANT FLOW:
Recruitment Details: VA primary care providers from 12 VA healthcare systems were enrolled and randomized to the intervention or control arm of the study. Veteran patients were subsequently recruited and enrolled into the study if they had an upcoming, scheduled appointment with a study provider. Veterans were automatically assigned to the study arm of the provider they were scheduled to see.
Groups:
- Intervention (MyPath): Providers were randomized to the intervention (MyPath) or usual care arm of the study. Patients scheduled to see providers randomized to this arm received a weblink to the MyPath decision tool via text message after study enrollment and prior to their scheduled visit.
- Usual Care Patients: Providers were randomized to the intervention (MyPath) or usual care arm of the study. Patients scheduled to see providers randomized to the usual care arm received no intervention text message and received usual care.
Period: Enrollment to Post-Visit - PATIENTS
Arm/Group | Intervention (MyPath) | Usual Care Patients
Started | 209 | 182
Completed | 190 | 159
Not Completed | 19 | 23
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Did not attend scheduled appointment with primary care provider | 16 | 18
Not completed — Pregnancy | 0 | 1
Period: 3-month Follow-up - PATIENTS
Arm/Group | Intervention (MyPath) | Usual Care Patients
Started | 190 | 159
Completed | 188 | 158
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1
Period: 6-month Follow-up - PATIENTS
Arm/Group | Intervention (MyPath) | Usual Care Patients
Started | 188 | 158
Completed | 184 | 156
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 2
Period: Enrollment to Post-Visit - PROVIDERS
Arm/Group | Intervention (MyPath) | Usual Care Patients
Started | 37 | 37
Completed | 34 | 32
Not Completed | 3 | 5
Not completed — No Veterans Enrolled in Study | 3 | 5

BASELINE CHARACTERISTICS:
Population: Per the study protocol, enrolled Veterans were excluded from the analytic sample if they were withdrawn from the study prior to any outcomes assessment due to non-attendance at their scheduled primary care visit, pregnancy diagnosed at the scheduled primary care visit, or self-withdrawal prior to outcomes assessment.
Groups:
- Intervention (MyPath) Patients: Patients scheduled to see providers randomized to this arm received a weblink to the MyPath decision tool via text message after study enrollment and prior to their scheduled visit.
- Usual Care Patients: Patients scheduled to see providers randomized to the usual care arm received no intervention text message and received usual care.
- Intervention (MyPath) Providers: This arm includes providers who were randomized to the intervention arm of the study and had at least one patient subsequently enroll.
- Usual Care Providers: This arm includes providers who were randomized to the usual care arm of the study and had at least one patient subsequently enroll.
- Total: Total of all reporting groups
Arm/Group | Intervention (MyPath) Patients | Usual Care Patients | Intervention (MyPath) Providers | Usual Care Providers | Total
Number analyzed (Participants) | 190 | 159 | 34 | 32 | 415
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 190 | 159 | 32 | 32 | 413
  >=65 years | 0 | 0 | 2 | 0 | 2
Age, Continuous [Mean (Full Range); unit: years of age] | 35.5 [21 to 45] | 35.1 [22 to 45] | 47.7 [29 to 67] | 47.7 [28 to 64] | 37.3 [21 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 159 | 32 | 29 | 410
  Male | 0 | 0 | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported Hispanic/Latina Ethnicity
  Participants
    Hispanic or Latino | 40 | 31 | 4 | 2 | 77
    Not Hispanic or Latino | 150 | 128 | 30 | 30 | 338
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported Racial Identity
  Participants
    American Indian or Alaska Native | 8 | 0 | 0 | 0 | 8
    Asian | 3 | 8 | 7 | 11 | 29
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 2
    Black or African American | 84 | 57 | 6 | 5 | 152
    White | 67 | 73 | 17 | 13 | 170
    More than one race | 12 | 7 | 1 | 0 | 20
    Unknown or Not Reported | 15 | 13 | 3 | 3 | 34
Sexual Orientation [Count of Participants; unit: Participants] — Self-reported sexual orientation identity. This question was asked of patients only (not providers).
  Participants
    Straight/Heterosexual | 149 | 120 | 0 | 0 | 269
    Lesbian/Gay | 14 | 14 | 0 | 0 | 28
    Bisexual/Pansexual | 22 | 19 | 0 | 0 | 41
    Other | 5 | 6 | 0 | 0 | 11
    Missing or Unknown | 0 | 0 | 34 | 32 | 66
Education [Count of Participants; unit: Participants] — Self-reported highest level of education. This was asked of patients only (not providers).
  Participants
    Some high school or GED | 17 | 11 | 0 | 0 | 28
    Some college or Associate's Degree | 81 | 61 | 0 | 0 | 142
    Bachelor's Degree or Higher | 91 | 87 | 0 | 0 | 178
    Missing or Unknown | 1 | 0 | 34 | 32 | 67
Health Insurance Status [Count of Participants; unit: Participants] — Self-reported whether patient has health insurance benefits separate/in addition to VA health coverage. This was asked of patients only (not providers).
  Participants
    Yes (separate health insurance) | 95 | 65 | 0 | 0 | 160
    No (VA coverage only) | 94 | 94 | 0 | 0 | 188
    Missing or Unknown | 1 | 0 | 34 | 32 | 67
Current thoughts/desires regarding pregnancy [Count of Participants; unit: Participants] — Self-report of patient's current thoughts/desires regarding pregnancy. This was asked of patients only (not providers).
  Participants
    Desires pregnancy now | 21 | 19 | 0 | 0 | 40
    Not trying to get pregnant, but okay with it | 23 | 27 | 0 | 0 | 50
    Not now, but desires pregnancy in future | 55 | 46 | 0 | 0 | 101
    Does not desire a future pregnancy (ever) | 60 | 45 | 0 | 0 | 105
    Unsure about pregnancy desires | 31 | 22 | 0 | 0 | 53
    Missing or Unknown | 0 | 0 | 34 | 32 | 66
Sex with a male partner, past 12 months [Count of Participants; unit: Participants] — Self-report of whether patient was sexually active with a male partner during the 12 months prior to enrollment. This was asked of patients only (not providers).
  Participants
    Yes | 147 | 117 | 0 | 0 | 264
    No | 43 | 41 | 0 | 0 | 84
    Missing or Unknown | 0 | 1 | 34 | 32 | 67
Participants enrolled per study provider [Mean (Full Range); unit: Veteran participants per provider] — Participants were included in the analytic sample if they attended a primary care visit at VA with a study provider.
  Veteran participants per provider | 5.6 [1 to 28] | 5.0 [1 to 18] | 5.6 [1 to 28] | 5.0 [1 to 18] | 5.3 [1 to 28]
Participants enrolled by study provider practice setting [Count of Participants; unit: Participants] — Some providers practice within a designated women's clinic at a VA Medical Center, while other study providers do not (i.e., practice in other general primary care clinics). Providers are categorized based on their own practice setting. Patients are categorized based on the practice setting of the provider they saw.
  Participants
    Women's clinic provider | 73 | 56 | 9 | 8 | 146
    Non-women's clinic provider | 117 | 103 | 25 | 24 | 269
Appointment modality [Count of Participants; unit: Participants] — Patients were included in the analytic sample if they attended a primary care visit at VA with a study provider. This measure captures whether the patient's visit was conducted in-person versus telehealth or virtual care. This is measured by self-report for patients who completed the post-visit survey. For patients who did not complete the post-visit survey, this was obtained through medical record review. This measure does not apply to providers.
  Participants
    In-person appointment | 156 | 122 | 0 | 0 | 278
    Virtual/telephone appointment | 34 | 37 | 0 | 0 | 71
    Does not apply (for providers) | 0 | 0 | 34 | 32 | 66
History of prior appointment(s) with study provider [Count of Participants; unit: Participants] — Patients were included in the analytic sample if they attended a primary care visit at VA with a study provider. This measure captures whether patient participants had medical record evidence of attending at last one prior appointment with their study provider within the 2 years prior to their study visit. This measure does not apply to study providers.
  Participants
    Yes (prior appointment(s) documented) | 135 | 136 | 0 | 0 | 271
    No (no prior appointment(s) documented) | 55 | 23 | 0 | 0 | 78
    Does not apply (providers) | 0 | 0 | 34 | 32 | 66
Annual household income [Count of Participants; unit: Participants] — Self-reported annual household income. This was asked of patients only (not providers).
  Participants
    <$20,000 | 9 | 9 | 0 | 0 | 18
    $20,000-$79,999 | 104 | 93 | 0 | 0 | 197
    >=$80,000 | 67 | 52 | 0 | 0 | 119
    Missing | 10 | 5 | 34 | 32 | 81
History of military deployment [Count of Participants; unit: Participants] — Self-reported measure of whether participant was ever deployed during their military service. This was asked of patients only (not providers).
  Participants
    Yes (deployed) | 108 | 80 | 0 | 0 | 188
    No (never deployed) | 81 | 79 | 0 | 0 | 160
    Missing | 1 | 0 | 34 | 32 | 67
History of military sexual trauma (MST) [Count of Participants; unit: Participants] — Obtained from patient VA medical records data (via the VA Corporate Data Warehouse). This captures whether a "yes" was every documented in the medical record for MST. This measure does not apply to providers.
  Participants
    Yes | 78 | 71 | 0 | 0 | 149
    No | 112 | 88 | 0 | 0 | 200
    Does not apply (providers) | 0 | 0 | 34 | 32 | 66
Ever experienced racial discrimination in VA care [Count of Participants; unit: Participants] — Measured using the Discrimination in Medical Settings Scale. Participants were prompted to think about care they have received from VA. Racial discrimination was defined as an answer of "sometimes," "most of the time," or "always" to any of the statements. This was asked of patients only (not providers).
  Participants
    Yes | 37 | 20 | 0 | 0 | 57
    No | 150 | 137 | 0 | 0 | 287
    Missing | 3 | 2 | 34 | 32 | 71
Satisfaction with VA care, past 12 months [Count of Participants; unit: Participants] — Measured using one question with answer options using a five-point scale ranging from "very satisfied' (score of 5) to "very dissatisfied" (score of 1). Overall satisfaction was defined as a score of 4 or 5 out of 5. This was asked of patients only (not providers).
  Participants
    Yes | 116 | 104 | 0 | 0 | 220
    No | 69 | 54 | 0 | 0 | 123
    Missing | 5 | 1 | 34 | 32 | 72
Has >=1 chronic medical condition (self-report) [Count of Participants; unit: Participants] — Veteran response (yes/no) to the following question: "Do you have any chronic medical conditions, such as diabetes, high blood pressure, migraines, asthma, or others?"
  Participants
    >=1 chronic medical condition | 131 | 110 | 0 | 0 | 241
    No chronic medical condition | 59 | 49 | 0 | 0 | 108
    Missing | 0 | 0 | 34 | 32 | 66
Has >=1 mental health condition (self-report) [Count of Participants; unit: Participants] — Veteran response (yes/no) to the following question: "Do you have any mental health conditions, such as depression, anxiety, bi-polar disorder, post-traumatic stress disorder, or others?" This was asked of patients only (not providers).
  Participants
    >=1 mental health condition | 158 | 140 | 0 | 0 | 298
    No mental health condition | 32 | 19 | 0 | 0 | 51
    Missing | 0 | 0 | 34 | 32 | 66
Provider Type [Count of Participants; unit: Participants] — Type of medical practitioner (self-report). This was asked of providers only (not patients).
  Participants
    Physician | 0 | 0 | 21 | 24 | 45
    Nurse Practitioner | 0 | 0 | 11 | 5 | 16
    Physician Assistant | 0 | 0 | 2 | 3 | 5
    Does not apply (patients) | 190 | 159 | 0 | 0 | 349
Years practicing in VA [Count of Participants; unit: Participants] — The number of years a provider has been practicing in VA. This was asked of providers only (not patients).
  Participants
    <5 years | 0 | 0 | 13 | 8 | 21
    5-10 years | 0 | 0 | 10 | 11 | 21
    >=10 years | 0 | 0 | 11 | 12 | 23
    Missing | 190 | 159 | 0 | 1 | 350

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Reproductive Needs Discussion With Shared Decision Making (SDM)
Description: Self-report of whether a discussion occurred during the scheduled primary care visit about pregnancy goals, prepregnancy health, or contraception that included shared decision making (SDM). SDM is measured by participant self-report with the CollaboRATE scale, which uses three 5-point Likert scale questions to assess SDM (score 0-12, with higher scores indicating more shared decision making; SDM defined using a top box score).
Time Frame: Within one month post-visit
Population: Enrolled Veterans were excluded from the analytic sample if they were withdrawn from the study prior to any outcomes assessment due to non-attendance at their scheduled primary care visit, pregnancy diagnosed at the scheduled primary care visit, or self-withdrawal prior to outcomes assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention (MyPath): Patients scheduled to see providers randomized to this arm received a weblink to the MyPath decision tool via text message after study enrollment and prior to their scheduled visit.
- Usual Care: Patients scheduled to see providers randomized to the usual care arm received no intervention text message and received usual care.
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 190 | 159
Participants
  Yes (discussion with SDM occurred) | 29 | 20
  No (discussion with SDM did not occur) | 139 | 119
  Missing (lost to follow-up for the post-visit survey) | 21 | 17
  Missing (declined to answer one or more outcome measure questions) | 1 | 3
Statistical Analysis 1: Comparison: Intervention (MyPath) vs Usual Care; We used a multilevel logistic regression model to test whether the outcome was significantly different in the intervention versus control arm. Analyses accounted for missing data in outcome and a priori adjustment variables through multiple imputation (MI) using Multiple Imputation by Chained Equations (MICE); Test type: Superiority; p = 0.31, Regression, Logistic — The threshold for significance was set at p<0.05; Model adjusted for site, provider clinic type, provider, Veteran age, Veteran race, Veteran education, and Veteran health insurance status; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.70 to 3.06]
Statistical Analysis 2: Comparison: Intervention (MyPath) vs Usual Care; Per the study protocol, to account for noncompliance, we estimated the "complier average causal effect" to estimate the causal effect of using the MyPath tool on the outcome. Our model accounted for missing data in outcome and baseline adjustment variables through multiple imputation (MI) using Multiple Imputation by Chained Equations (MICE) in R; Test type: Superiority; Regression, Logistic — Threshold for significance was set at p<0.05; [statistical method as in outcome 1, analysis 1]; P-value and estimated OR (95% CI) is not available because the model did not converge

2. Secondary Outcome: Occurrence of Reproductive Needs Discussion
Description: Self-report of whether a discussion of pregnancy goals, prepregnancy health, or contraception occurred during the scheduled primary care visit, regardless of occurrence of SDM.
Time Frame: Within one month post-visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 190 | 159
Participants
  Yes (discussion occurred) | 119 | 93
  No (discussion did not occur) | 49 | 49
  Missing (lost to follow-up for post-visit survey) | 21 | 17
  Missing (declined one or more measure questions) | 1 | 0
Statistical Analysis 1: Comparison: Intervention (MyPath) vs Usual Care; We used a multilevel logistic regression model to test whether the outcome was significantly different in the intervention versus control arm, using an Intent to Treat approach. Analyses accounted for missing data in outcome and baseline adjustment variables through multiple imputation (MI) using Multiple Imputation by Chained Equations (MICE); Test type: Superiority; p = 0.26, Regression, Logistic — Threshold for significance was set at p<0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.79 to 2.38]
Statistical Analysis 2: Comparison: Intervention (MyPath) vs Usual Care; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.019, Regression, Logistic — Threshold for significance was set at p<0.05; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.46, 95% CI 2-sided [1.23 to 9.76]

3. Secondary Outcome: Perceived Self-efficacy in Communicating With Providers
Description: Assessed with a modified version of the validated 5-item Perceived Efficacy in Patient-Provider Interactions (PEPPI) scale, which uses five Likert scale questions ranging from 1 to 5 (score 5-25, with higher scores indicating higher levels of perceived efficacy).
Time Frame: Within one month post-visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 190 | 159
Score | 19.8 (4.8) | 20.6 (4.4)
Statistical Analysis 1: Comparison: Intervention (MyPath) vs Usual Care; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.27, Regression, Linear — Threshold for significance was set at p<0.05; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -0.62, 95% CI 2-sided [-1.71 to 0.48]
Statistical Analysis 2: Comparison: Intervention (MyPath) vs Usual Care; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.42, Regression, Linear — Threshold for significance was set at p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-2.91 to 1.22]

4. Secondary Outcome: Reproductive Health Knowledge
Description: Participant responses to 14 items assessing knowledge of fertility, prepregnancy health, and contraception. The measure is self-developed and derived from previously published assessments of fertility and contraceptive knowledge. Responses will be coded as correct vs. incorrect, with "don't know" coded as incorrect (score 0-14, with higher scores indicating more accurate knowledge).
Time Frame: Within one month post-visit
Population: This outcome was measured within a prespecified analytic subgroup (n=150) defined at study enrollment (pre-intervention) as potentially at risk of unintended pregnancies, defined using baseline measures of current pregnancy desires (does not desire pregnancy now or within the next year), pregnancy capability (does not report a prior tubal sterilization) and sexual activity (reports sex with a male partner in the past 12 months).
Measure: Mean (Standard Deviation); unit: Number correct
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Number correct | 7.94 (2.64) | 7.89 (2.36)
Statistical Analysis 1: Comparison: Intervention (MyPath) vs Usual Care; We used a multilevel logistic regression model to test whether the outcome was significantly different in the intervention versus control arm, using an Intent to Treat approach; Test type: Superiority; p = 0.45, Regression, Linear — Threshold for significance was set at p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.35, 95% CI 2-sided [-0.56 to 1.26]
Statistical Analysis 2: Comparison: Intervention (MyPath) vs Usual Care; Per the study protocol, to account for noncompliance, we estimated the "complier average causal effect" to estimate the causal effect of using the MyPath tool on the outcome; Test type: Superiority; p = 0.09, Regression, Linear — Threshold for significance was set at p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [-0.15 to 2.02]

5. Secondary Outcome: Contraceptive Decision Conflict
Description: Assessed with the Decision Conflict Scale (DCS), a validated measure to assess patients' decisional conflict in medical decision making. The DCS includes 16-items with 5-point Likert scale response options ranging from 0-4. Scores are converted to range from 0 (no decisional conflict) to 100 (highest decisional conflict). This measure will be obtained in a pre-defined subset of participants at risk of unintended pregnancy.
Time Frame: Within one month post-visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Score | 16.94 (17.57) | 20.04 (20.67)
Statistical Analysis 1: Comparison: Intervention (MyPath) vs Usual Care; We used a multilevel regression model to test whether the outcome was significantly different in the intervention versus control arm, using an Intent to Treat approach; Test type: Superiority; p = 0.56, Regression, Linear — Threshold for significance was set at p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.26, 95% CI 2-sided [-9.94 to 5.42]
Statistical Analysis 2: Comparison: Intervention (MyPath) vs Usual Care; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.02, Regression, Linear — Threshold for significance was set at p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.72, 95% CI 2-sided [-25.37 to -2.06]

6. Secondary Outcome: Confidence That Contraceptive Method is "Right for me."
Description: Assessed using a single question ("How confident are you that this contraceptive method is right for you?") with Likert response options from 1 (not at all confident) to 5 (completely confident). This measure will be obtained in a pre-defined subset of participants at risk of unintended pregnancy.
Time Frame: Within one month post-visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Scores on a scale | 4.29 (1.05) | 4.29 (1.06)
Statistical Analysis 1: Comparison: Intervention (MyPath) vs Usual Care; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.84, Regression, Linear — Threshold for significance was set at p<0.05; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.38 to 0.47]
Statistical Analysis 2: Comparison: Intervention (MyPath) vs Usual Care; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.27, Regression, Linear — Threshold for significance was set at p<0.05; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [-0.35 to 1.25]

7. Secondary Outcome: Choice of Prescription or Procedural Contraceptive Method
Description: Self-report of continuing or changing to a prescription or procedural method after their visit. Prescription or procedural methods are defined as any of the following: birth control pills, patch, ring, injection, implants, IUDs, and male and female sterilization. This measure will be obtained in a pre-defined subset of participants at risk of unintended pregnancy.
Time Frame: Within one month post-visit
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Participants
  Prescription or procedural method | 52 | 35
  Non-prescription or no method | 25 | 17
  Missing (lost to follow-up) | 7 | 10
  Missing (did not answer question(s)) | 2 | 2

8. Secondary Outcome: Choice of Procedural Contraceptive Method
Description: Self-report of continuing or changing to a procedural method after their visit. Procedural methods are defined as any of the following: implants, IUDs, and male and female sterilization. This measure will be obtained in a pre-defined subset of participants at risk of unintended pregnancy.
Time Frame: Within one month post-visit
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Participants
  Procedural method | 28 | 20
  Non-procedural or no method | 49 | 32
  Missing (lost to follow-up for post-visit survey) | 7 | 10
  Missing (did not answer question(s)) | 2 | 2

9. Secondary Outcome: Use of Prescription or Procedural Contraceptive Method
Description: Self-reported use of a prescription or procedural method at follow-up. Prescription or procedural methods are defined as any of the following: birth control pills, patch, ring, injection, implants, IUDs, and male and female sterilization. This measure will be obtained in a pre-defined subset of participants at risk of unintended pregnancy.
Time Frame: 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Participants
  Prescription or procedural method | 41 | 28
  Non-prescription or no method | 23 | 14
  Missing (lost to follow-up 6-month survey) | 22 | 21
  Missing (did not answer question(s) due to pregnancy) | 0 | 1

10. Secondary Outcome: Use of Procedural Contraceptive Method
Description: Self-reported use of a procedural method at follow-up. Procedural methods are defined as any of the following: implants, IUDs, and male and female sterilization. This measure will be obtained in a pre-defined subset of participants at risk of unintended pregnancy.
Time Frame: 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Participants
  Procedural method | 22 | 17
  Non-procedural or no method | 42 | 25
  Missing (lost to follow-up 6-month survey) | 22 | 21
  Missing (did not answer question(s) due to pregnancy) | 0 | 1

11. Secondary Outcome: Continuous Use of Any Contraception
Description: Self-reported use of a contraceptive method over the past 6 months without a gap of greater than 4 weeks. This combines self-reported use at 3 months and 6 months. This measure will be obtained in a pre-defined subset of participants at risk of unintended pregnancy. For participants lost to follow-up at the 6 month timepoint, their 6-month values will be singly imputed, carrying forward 3-month continuous use reports when those data are available.
Time Frame: 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Participants
  Continuous use over 6 months | 62 | 46
  Non-continuous use over 6 months | 13 | 6
  Missing (lost to follow-up for 6 month survey) | 11 | 11
  Missing (did not answer question(s) due to pregnancy) | 0 | 1

12. Secondary Outcome: Continuous Use of Prescription or Procedural Contraception
Description: Self-reported use of a prescription or procedural contraceptive method over the past 6 months without a gap of greater than 4 weeks. Prescription or procedural methods are defined as any of the following: birth control pills, patch, ring, injection, implants, IUDs, and male and female sterilization. This measure will be obtained in a pre-defined subset of participants at risk of unintended pregnancy.
Time Frame: 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Participants
  Continuous Use of Rx/Procedural Contraception | 45 | 31
  Non-Continuous Use of Rx/Procedural Contraception | 30 | 21
  Missing (lost to follow-up for 6-month survey) | 11 | 11
  Missing (did not answer question(s) due to pregnancy) | 0 | 1

13. Secondary Outcome: Continuous Use of Procedural Contraception
Description: Self-reported use of a procedural contraceptive method over the past 6 months without a gap of greater than 4 weeks. Procedural methods are defined as any of the following: implants, IUDs, and male and female sterilization. This measure will be obtained in a pre-defined subset of participants at risk of unintended pregnancy.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Participants
  Continuous Use of Procedural Contraception | 27 | 19
  Non-continuous Use of Procedural Contraception | 48 | 33
  Missing (lost to follow-up for 6-month survey) | 11 | 11
  Missing (did not answer question(s) due to pregnancy) | 0 | 1

14. Secondary Outcome: Contraceptive Method Satisfaction
Description: Assessed using a single question ("How satisfied are you with your current birth control method") with Likert response options from 1 (very dissatisfied) to 5 (very satisfied). This measure will be obtained in a pre-defined subset of participants at risk of unintended pregnancy. While this outcome was measured at 6 months, for participants lost to follow-up at 6 months, we singly imputed these data by pulling forward their 3-month satisfaction, when available.
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Score | 4.28 (1.01) | 4.35 (0.95)

15. Secondary Outcome: Incidence of Unplanned Pregnancy
Description: Proportion of participants who self-report an unplanned pregnancy, as determined by responses to the 6-item London Measure of Unplanned Pregnancy. The London Measure includes items measuring attitude towards an experienced pregnancy and behaviors before pregnancy to determine the intendedness of pregnancy. The score range of the London Measure is 0-12, with a score of <10 indicating unplanned pregnancy and a score of 10 or higher indicating planned pregnancy. This measure will be obtained in a pre-defined subset of participants at risk of unintended pregnancy.
Time Frame: 6 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Participants
  Unplanned pregnancy | 0 | 1
  No unplanned pregnancy | 64 | 42
  Missing (lost to follow-up 6 month survey) | 22 | 21

16. Secondary Outcome: Confidence That Current Contraceptive Method is "Right for me."
Description: as for outcome 6
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Scores on a scale | 4.26 (0.90) | 4.21 (0.98)

17. Other Pre Specified Outcome: Goals-concordant Contraceptive Use
Description: Self-reported contraception use among participants at 6 months that is consistent with their orientation towards pregnancy at 6-months (desires pregnancy now, not trying but OK with it, desires pregnancy later but not now, never desires pregnancy, not sure), regardless of their intention at baseline. This measure will be obtained in a pre-defined subset of participants at risk of unintended pregnancy. For Veterans who desire pregnancy now, goals-concordant contraceptive use is defined as not using contraception. For Veterans who desire pregnancy later, never, or are unsure, goals-concordant contraceptive use is defined as using contraception. For Veterans who are not trying to get pregnant but would be OK with it, goals-concordant contraceptive use is defined as either using or not using contraception.
Time Frame: 6 months
Population: This outcome was measured within a prespecified analytic subgroup (n=150) defined at study enrollment (pre-intervention) as potentially at risk of unintended pregnancies, defined using baseline measures of pregnancy desires (does not desire pregnancy now or within the next year), pregnancy capability (does not report a prior tubal sterilization) and sexual activity (reports sex with a male partner in the past 12 months).
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Participants
  Yes (goals-concordant contraceptive use) | 50 | 38
  No (not goals-concordant contraceptive use) | 14 | 4
  Missing (lost to follow-up at 6-months) | 22 | 21
  Missing (not asked question(s) due to pregnancy) | 0 | 1

18. Other Pre Specified Outcome: Contraceptive Knowledge
Description: Participant responses to 8 items assessing knowledge of contraception. The measure derived from previously published assessments of contraceptive knowledge. Responses will be coded as correct vs. incorrect, with "don't know" coded as incorrect (score 0-8, with higher scores indicating more accurate knowledge).
Time Frame: Within one month post-visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Intervention (MyPath) | Usual Care
Number analyzed (Participants) | 86 | 64
Score | 4.42 (1.72) | 4.15 (1.54)
Statistical Analysis 1: Comparison: Intervention (MyPath) vs Usual Care; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.21, Regression, Linear — threshold for significance set at <0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.22 to 0.99]
Statistical Analysis 2: Comparison: Intervention (MyPath) vs Usual Care; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.04, Regression, Linear — Threshold for significance was set at p<0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.89, 95% CI [0.04 to 1.75]

ADVERSE EVENTS:
Time Frame: from enrollment through 6 months follow-up
Groups:
- Intervention (MyPath) Patients: Patients scheduled to see providers randomized to the intervention arm received a weblink to the MyPath decision tool via text message after study enrollment and prior to their scheduled visit.
- Intervention (MyPath) Providers: Providers randomized to the intervention arm.
- Usual Care Providers: Providers randomized to the usual care arm.
Arm/Group | Intervention (MyPath) Patients | Usual Care Patients | Intervention (MyPath) Providers | Usual Care Providers
All-Cause Mortality (participants affected / at risk) | 0/209 | 0/182 | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/209 | 0/182 | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/209 | 0/182 | 0/37 | 0/37

LIMITATIONS AND CAVEATS:
Limitations of the study that impacted our ability to assess the effectiveness of the intervention include (1) lower than expected adherence (use of the MyPath tool) and (2) higher than expected lost-to-follow-up for our primary outcome at the post-visit timeframe.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT04584294/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT04584294/ICF_000.pdf